CLINICAL TRIAL: NCT03608020
Title: A Safety Lead-In/Randomized Phase 2 Study of BMX-001 as a Therapeutic Agent for Treatment of Cancer Patients With Multiple Brain Metastases Undergoing Whole-Brain Radiotherapy
Brief Title: A Trial for Treatment of Cancer Patients With Multiple Brain Metastases Undergoing Whole-Brain Radiotherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Cessation of grant funding
Sponsor: BioMimetix JV, LLC (Industry)
Collaborators: Duke Cancer Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMX-MBM-001; 1R44CA228694-01 (NIH)
Record Dates: First submitted 2018-06-14; First posted 2018-07-31 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Multiple Brain Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WBRT + BMX-001 (Active Comparator): Whole brain radiation therapy in combination with BMX-001 (subcutaneous injection of 28 mg loading dose, followed by subsequent 14 mg twice per week for 2 weeks).
  Interventions: Drug: BMX-001; Radiation: Whole Brain Radiation Therapy
- Whole Brain Radiation Therapy (No Intervention): Whole brain radiation therapy per standard of care.

INTERVENTIONS:
Drug: BMX-001 — Manganese butoxyethyl pyridyl porphyrin
  Other Names: Whole Brain Radiation Therapy
  Arms: WBRT + BMX-001
Radiation: Whole Brain Radiation Therapy — Whole Brain Radiation Therapy per standard of care.
  Arms: WBRT + BMX-001

SUMMARY:
This protocol is for a lead-in safety study of 5 patients followed by a randomized Phase 2 clinical trial of BMX-001, a new class of pharmaceutical, in 64 patients with multiple brain metastases (MBM) undergoing whole brain radiation therapy (WBRT). Preliminary studies have demonstrated that BMX-001 provides protection of normal tissues from radiation-induced injury and augments tumor growth inhibition.

DETAILED DESCRIPTION:
This protocol is for a Phase 1 safety lead-in clinical trial of BMX-001 in combination with WBRT in 5 patients with MBM. Demonstrating safety of the selected MTD of BMX-001 in patients with MBM undergoing standard protocol WBRT will be the "go/no-go" criteria for proceeding to Phase 2.

Phase 2 is a randomized open-label Phase 2 clinical trial of 64 patients with MBM, half receiving BMX-001 in combination with WBRT and half receiving WBRT alone.

Subjects are treated with BMX-001 for a total of 19 days, during which time they receive radiation therapy. Following completion of radiation therapy, subjects will be followed for an additional one year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed diagnosis of a non-small cell lung cancer, breast cancer, melanoma or renal cell cancer primary
* Subjects must have >5 contrast-enhancing lesions, never previously treated with SRS and/or surgical resection, on a contrast-enhanced T1-weighted brain MRI performed within two weeks of enrollment, with at least one lesion >0.5cm in greatest dimension
* Physical examination by a radiation oncologist or medical oncologist within 14 days of the start of WBRT
* Plan to be treated with WBRT to a dose of 30 Gy in 10 fractions
* Age * 18 years
* Karnofsky Performance Status (KPS) ≥ 70
* Hemoglobin ≥ 9.0 g/dl, ANC ≥ 1,500 cells/*l, platelets ≥ 125,000 cells/*l
* Serum creatinine ≤ 1.5 mg/dl, serum SGOT and bilirubin ≤ 1.5 times upper limit of normal
* Signed informed consent approved by the Institutional Review Board
* If sexually active, patients must agree to use appropriate contraceptive measures for the duration of the study and for 6 months afterwards as stated in the informed consent
* Able to provide study specific informed consent
* Willing to follow study procedures, complete QOL questionnaires and neurocognitive testing as described in the protocol
* Negative serum pregnancy test for women of child bearing potential within 48 hours of first dose of BMX

Exclusion Criteria:

* Active infection requiring IV antibiotics 7 days before enrollment
* Hypertension requiring 3 or more anti-hypertensive medications to control
* Requirement for concurrent treatment with nitrates or other drugs that may, in the judgment of the treating investigator, create a risk for a precipitous decrease in blood pressure
* History of syncope within the last 6 months
* Subjects receiving prohibited medications listed in Section 6.4.2 of this protocol are not eligible. Subjects who can safely stop taking a prohibited medication at least 7 days prior to the first dose of BMX may participate at the discretion of the treating physician.
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* Women who are breast feeding
* Known hypersensitivity to compounds of similar chemical composition to BMX-001
* Prior surgical resection for brain metastases and/or stereotactic radiosurgery for up to 5 brain metastases in total are permitted if performed at least 1 month prior to planned WBRT under this protocol.
* Prior whole brain radiation therapy
* Patients with diffuse leptomeningeal disease (carcinomatous meningitis)
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >480 milliseconds (ms) (CTCAE grade 1)
* A history of additional risk factors for TdP (e.g., congestive heart failure, hypokalemia, known family history of Long QT Syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Assess safety and tolerability of WBRT + BMX-001 through proportion of patients who experience grade 4 or 5 study drug related adverse events. | 1 year
  AEs will be assessed according to the CTCAE version 5.0. If CTCAE grading does not exist for an AE, the severity of the AE will be graded as mild (1), moderate (2), severe (3), life-threatening (4), or fatal (5). Initially 5 patients will be accrued and treated with WBRT + BMX-001 as a lead-in safety phase. Enrollment to the randomized phase of the study will not proceed if patients in the safety lead-in phase experience the following:
  * Two or more patients are unable to complete radiation therapy (RT) due to toxicity related to BMX-001 (alone or in combination with RT.
  * Two or more patients experience delay in starting RT due to toxicity related to BMX-001 (alone or in combination with RT).
  If any patient experiences a grade 4 or 5 BMX-001-related adverse event within Arm A (WBRT + BMX-001), accrual will be suspended and the experience of the patient will be carefully reviewed by the clinical team and the study's DSMB.
Compare neurocognition in WBRT + BMX-001 vs. WBRT alone using cumulative score of HVLT-R, TMT A&B and COWA over time. | 1 Year
  Subjects will complete three standardized tests (Hopkins Verbal Learning Test - Revised, Trail Making Test A&B, and Controlled Oral Word Association test) at baseline, 1 month after completion of WBRT and every 3 months after completion of WBRT. The cumulative score of these three tests will be used to assess change.

SECONDARY OUTCOMES:
Compare survival in WBRT + BMX-001 vs WBRT alone | 1 Year
  Survival
Compare local recurrence rate in WBRT + BMX-001 vs WBRT alone | 1 Year
  Median time to local brain failure or progression
Compare distant brain failure rate in WBRT + BMX-001 vs WBRT alone | 1 Year
  Median time to distant brain failure
Compare rate of neurologic death in WBRT + BMX-001 vs WBRT alone | 1 Year
  Proportion of patients who are dead within 1 year of initiation of WBRT due to neurologic disease and/or disseminated leptomeningeal carcinomatosis.

OTHER OUTCOMES:
Compare rate of radionecrosis in WBRT + BMX-001 vs WBRT alone | 1 Year
  Proportion of patients with enlarged and/or symptomatic brain lesions with no viable tumor on biopsy
Compare QoL in WBRT + BMX-001 vs WBRT alone | 1 Year
  Mean change from baseline at each follow-up assessment

CONTACTS AND LOCATIONS:
Overall Officials: John Kirkpatrick, MD, Principal Investigator — Duke Cancer Institute
Locations (4):
- United States (4):
  - University of Kentucky, Lexington, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - Duke Cancer Institute, Durham, North Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No